CLINICAL TRIAL: NCT00296595
Title: Physiological Mechanisms Underlying the Effects of PUFA and Antioxidants on Postprandial Lipemia, Oxidative Stress, Endothelial Dysfunction and Inflammation in Men
Brief Title: Effects of n-3 Polyunsaturated Fatty Acids and Antioxidants on Postprandial Hyperlipidemia and Vascular Function in Men
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Charles Couillard, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOP-64438
Record Dates: First submitted 2006-02-09; First posted 2006-02-27 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Cardiovascular Diseases; Vasodilation
MeSH Terms: conditions — Cardiovascular Diseases; Aneurysm | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Placebo capsules + 500 mL/day of placebo juice
  Interventions: Behavioral: Nutrition
- Cranberry Juice (Experimental): Placebo capsules + 500 mL/day of cranberry juice
  Interventions: Behavioral: Nutrition
- Fish Oil (Experimental): 2 g/day of fish oil + 500 mL/day of placebo juice
  Interventions: Behavioral: Nutrition
- Cranberry Juice + Fish Oil (Experimental): 2 g/day of fish oil + 500 mL/day of cranberry juice
  Interventions: Behavioral: Nutrition

INTERVENTIONS:
Behavioral: Nutrition

SUMMARY:
Diet has long been used as a way to provide enough nutrients to an individual in order to meet metabolic requirements. However, recent scientific advancements have suggested that beyond meeting nutrition needs, diet may also be health promoting through the modulation of various body functions. In a way, the role of nutrition has evolved from hunger satisfaction and maintenance of body integrity to the promotion of a state of well-being and prevention of important chronic diseases such as cancer, diabetes and cardiovascular disease (CVD). In recent years, n-3 polyunsaturated fatty acids (PUFA) have attracted much attention as consumption of a n-3 PUFA rich diet has been reported to reduce CVD risk. However, n-3 PUFA are also highly susceptible to free radical damage and therefore could be unable to fully exert their health benefits under an oxidative stress condition. The general objective of the present application is to investigate the mechanisms by which n-3 PUFA improve cardiovascular health in abdominal obesity and explore the potential of dietary antioxidants to modulate these effects in individuals at high risk of oxidative stress. For that purpose, we plan to study the changes in fasting and postprandial plasma lipoprotein-lipid levels, markers of lipid and lipoprotein oxidation, inflammation and endothelial dysfunction following 12 weeks of n-3 PUFA supplementation with or without low-calorie cranberry juice cocktail (as a source of antioxidants) in a group of 160 men. We feel that the present study will broaden our understanding of the physiological mechanisms underlying the beneficial effects of consuming unsaturated fatty acids and give further insights on the role of antioxidants in preserving and potentiating these cardiovascular health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference > 90 cm
* Fasting triglycerides > 1.7 mmol/L
* No use (ever) of medications for the treatment for dyslipidemia or hypertension

Exclusion Criteria:

* Alcohol consumption > 1 drink per day i.e ~15 g of alcohol/day or the equivalent of 1 beer (12 oz or 341 mL), 1 glass of wine (4 oz or 125 mL) or 1 ounce (30 mL) of liquor.
* Chronic use of supplements (vitamins, minerals or flavonoids)
* Body mass index > 35 kg/m2
* Chronic diseases: CHD, diabetes, etc.
* Smokers (1 or more cigarette/day)
* Dyslipidemia secondary to renal insufficiency, hypothyroidism or others
* Any prior or current use of medications known to affect lipoprotein-lipid metabolism (e.g. statins, fibrates), endothelial function (hypotensive drugs). Use (ever) of anticoagulant drugs (e.g. warfarin) because of possible detrimental interaction with the consumption of cranberry juice. Current or recent (<2 weeks) use of anti-inflammatory drugs Note: If for any reason, a subject would have to go an any of these drugs during the protocol, they would be automatically dropped from the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in postprandial lipemia, oxidative stress, endothelial activation and inflammation: TG (plasma, chylomicron and VLDL), OxLDL, 8-iso-PGF2alpha, ICAM-1, VCAM-1, E-selectin and CRP concentrations | June 2008

SECONDARY OUTCOMES:
Changes in arterial flow-mediated vasodilatory response | June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Charles Couillard, Ph.D., Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceuticals and Functional Foods, Québec, Quebec, Canada

REFERENCES:
- [Background] Ruel G, Pomerleau S, Couture P, Lamarche B, Couillard C. Changes in plasma antioxidant capacity and oxidized low-density lipoprotein levels in men after short-term cranberry juice consumption. Metabolism. 2005 Jul;54(7):856-61. doi: 10.1016/j.metabol.2005.01.031. PMID 15988692
- [Background] Couillard C, Ruel G, Archer WR, Pomerleau S, Bergeron J, Couture P, Lamarche B, Bergeron N. Circulating levels of oxidative stress markers and endothelial adhesion molecules in men with abdominal obesity. J Clin Endocrinol Metab. 2005 Dec;90(12):6454-9. doi: 10.1210/jc.2004-2438. Epub 2005 Sep 27. PMID 16189262